CLINICAL TRIAL: NCT01885689
Title: Phase II Study of Clofarabine and High-Dose Melphalan Conditioning Prior to Allogeneic Hematopoietic Cell Transplantation for Myelodysplasia or Acute Leukemia in Remission
Brief Title: Clofarabine and Melphalan Before Donor Stem Cell Transplant in Treating Patients With Myelodysplasia, Acute Leukemia in Remission, or Chronic Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13130; NCI-2013-01193 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2023-04-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia in Remission; Myelodysplastic Syndrome; Secondary Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Clofarabine; Melphalan; Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (clofarabine, melphalan, transplant) (Experimental): CONDITIONING REGIMEN: Patients receive clofarabine IV over 2 hours on days -9 to -5 and melphalan IV over 30 minutes on day -4.
  TRANSPLANT: Patients undergo allogeneic hematopoietic stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Beginning on day -3, patients receive tacrolimus IV or PO and sirolimus PO once daily with taper per City of Hope standard operating procedure.
  Interventions: Drug: clofarabine; Drug: melphalan; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: tacrolimus; Drug: sirolimus; Other: Pharmacological Study

INTERVENTIONS:
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic hematopoietic stem cell transplant
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well clofarabine and melphalan before a donor stem cell transplant works in treating patients with a decrease in or disappearance of signs and symptoms of myelodysplasia or acute leukemia (disease is in remission), or chronic myelomonocytic leukemia. Giving chemotherapy, such as clofarabine and melphalan, before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into a patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving clofarabine and melphalan before transplant may help prevent the cancer from coming back after transplant, and they may cause fewer side effects than standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Following a patient safety lead-in, determine the anti-tumor activity of clofarabine given in combination with high-dose melphalan as assessed by 2-year progression-free survival (PFS).

II. Estimate overall survival (OS), cumulative incidence (CI) of relapse/progression and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

III. Summarize toxicities/complications by organ and severity, including acute and chronic graft-vs-host disease (GVHD), and infection.

OUTLINE:

CONDITIONING REGIMEN: Patients receive clofarabine intravenously (IV) over 2 hours on days -9 to -5 and melphalan IV over 30 minutes on day -4.

TRANSPLANT: Patients undergo allogeneic hematopoietic stem cell transplant on day 0.

GVHD PROPHYLAXIS: Beginning on day -3, patients receive tacrolimus IV or orally (PO) and sirolimus PO once daily with taper per City of Hope standard operating procedure.

After completion of study treatment, patients are followed up once weekly for 60 days, at 100, and 180 days, at one year, and then yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients in 1st or 2nd remission with acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL), who are eligible for stem cell transplant. Remission defined as no circulating blasts, < 5% blasts in the bone marrow, normalization of previously detected cytogenetic abnormalities, no extramedullary disease
* High risk myelodysplastic syndrome (MDS)

  * Intermediate II and high risk by International Prognostic Scoring System (IPSS)
  * Intermediate, high, or very high by World Health Organization (WHO) classification-based Prognostic Scoring System (WPSS)
  * Transfusion dependent
  * Therapy-related MDS or MDS evolved from previous hematological disorder (excepting myelofibrosis)
* Patients with chronic myelomonocytic leukemia (CMML) are allowed to be enrolled
* Patients with MDS that has evolved to AML must be in remission
* Patients must not be eligible for full ablative regimens by the attending physician
* Patients with AML or MDS arising from myeloproliferative neoplasm can be enrolled after principal investigator (PI) approval on case to case basis, depends on the spleen size and degree of bone marrow fibrosis
* Performance status of >= 70% on the Karnofsky scale
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect she is pregnant while participating on the trial, she should inform her treating physician immediately
* Bone marrow and peripheral blood studies must be available for confirmation of diagnosis; cytogenetics, flow cytometry, and molecular studies (such as Flt-3 status) will be obtained as per standard practice
* Bone marrow aspirates/biopsies should be performed within 28 (+ 4 day window) days from registration to confirm disease remission status
* A pretreatment measured creatinine clearance (absolute value) of >= 60 mL/minute
* Patients must have a serum bilirubin =< 2.0 mg/dl
* Patients must have serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 2.5 times the institutional upper limit of normal
* Ejection fraction measured by echocardiogram or multi gated acquisition scan (MUGA) > 50%
* Diffusing capacity of the lung for carbon monoxide (DLCO) or forced expiratory volume in 1 second (FEV1) > 45% predicted
* Availability of a human leukocyte antigen (HLA) matched (6/6) sibling donor or 8/8 matched unrelated donor; Donors with mismatch at HLA-A, HLA-B, HLA-C, and HLA-DR will be reviewed by matched unrelated donor (MUD) committee and allowed if their mismatch with the recipient does not require additional GVHD prophylaxis (other than tacrolimus and sirolimus), donors with mismatch at HLA-DQ or HLA-DPB are eligible; donor evaluation according to City of Hope (COH) standard operating procedure (SOP)
* Donor stem cell source can be either peripheral blood or bone marrow
* All patients must have a psychosocial evaluation prior to transplant as per COH SOP
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* ALL or AML patients who received chemotherapy (induction or consolidation) can proceed to transplant once bone marrow cellularity is > 10 % with no evidence of leukemia

Exclusion Criteria:

* Patients who have received a prior autologous or allogeneic transplant are excluded
* Patients with significant hepatic dysfunction (not meeting liver function tests [LFT] eligibility criteria)
* Patients with MDS evolved into AML that is not in remission
* Patients with acute promyelocytic leukemia
* Patients with myeloproliferative neoplasms
* Patients with suspected or proven central nervous system (CNS) leukemia; (diagnostic lumbar puncture not required before enrollment)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active or poorly controlled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and lactating women are excluded from this study
* Patients who do not agree to practice effective forms of contraception
* Human immunodeficiency virus (HIV)-positive patients are excluded from this study
* Patients are excluded if they are hepatitis B surface antigen (sAg), hepatitis B (Hep B) core antibody (cAb), or hepatitis C (Hep C) positive. Patients with Hepatitis B cAB positive and Hepatitis B PCR negative are eligible if they started prophylactic treatment prior to registration to trial
* Patients who have received radiation therapy as part of their leukemia treatment may be ineligible and individual cases must be presented to the study principal investigator (PI) for determination of eligibility
* Any psychiatric, social or compliance issues that, in the treating physician's opinion, will interfere with completion of the transplant treatment and follow up
* Medical or psychiatric reasons which make the donor unlikely to tolerate or cooperate with filgrastim (G-CSF) therapy or leukapheresis or bone marrow harvest
* Known allergies to clofarabine, melphalan, sirolimus or tacrolimus
* Patients with other active malignancies (besides AML, ALL, MDS) requiring treatment or where there is concern of progression are ineligible for this study; however, patients with previously treated skin cancer, early stage cervical or prostate cancer may be eligible if there is no evidence of residual disease
* Cord blood as a donor source is not acceptable
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2026-09-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Monzr Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 patients consented to the study. 52 of them became eligible and received the study treatment.
Groups:
- Treatment (Clofarabine, Melphalan, Transplant): CONDITIONING REGIMEN: Patients receive clofarabine IV over 2 hours on days -9 to -5 and melphalan IV over 30 minutes on day -4.
  TRANSPLANT: Patients undergo allogeneic hematopoietic stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Beginning on day -3, patients receive tacrolimus IV or PO and sirolimus PO once daily with taper per City of Hope standard operating procedure.
  clofarabine: Given IV
  melphalan: Given IV
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic hematopoietic stem cell transplant
  tacrolimus: Given IV or PO
  sirolimus: Given PO
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Clofarabine, Melphalan, Transplant)
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Clofarabine, Melphalan, Transplant)
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 2 Years
Description: Progression-free survival (PFS) is defined as time from start of protocol treatment to disease relapse/progression, death or last contact, whichever occurs first. Progression-free survival was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula.
Time Frame: From start of protocol treatment to death due to any cause, disease relapse/progression, or last follow-up, whichever comes first, assessed up to 2 years.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Treatment (Clofarabine, Melphalan, Transplant)
Number analyzed (Participants) | 52
percent probability | 54 [39 to 66]

2. Secondary Outcome: Overall Survival at 2 Years
Description: Overall survival (OS) is defined as time from start of protocol treatment to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula.
Time Frame: From start of protocol treatment to death due to any cause, or last follow-up, whichever comes first, assessed up to 2 years.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Treatment (Clofarabine, Melphalan, Transplant)
Number analyzed (Participants) | 52
percent probability | 67 [53 to 78]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to Day 100 post-transplant. All-Cause Mortality was assessed from start of protocol treatment to death due to any cause, or last follow-up, whichever comes first, assessed up to 6 years.
Arm/Group | Treatment (Clofarabine, Melphalan, Transplant)
All-Cause Mortality (participants affected / at risk) | 23/52
Serious Adverse Events (participants affected / at risk) | 16/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Clofarabine, Melphalan, Transplant) (N=52)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3)
Lung infection (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 3 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Clofarabine, Melphalan, Transplant) (N=52)
Anemia (Blood and lymphatic system disorders) | 51 (118)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 31 (34)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrial flutter (Cardiac disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 12 (17)
Chest pain - cardiac (Cardiac disorders) | 6 (6)
Heart failure (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 18 (24)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 2 (3)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 7 (9)
Eye pain (Eye disorders) | 3 (3)
Floaters (Eye disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 36 (55)
Anal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 14 (16)
Colitis (Gastrointestinal disorders) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Colonic ulcer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 22 (27)
Diarrhea (Gastrointestinal disorders) | 51 (87)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 4 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (8)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 23 (44)
Hemorrhoids (Gastrointestinal disorders) | 6 (7)
Ileus (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 29 (37)
Nausea (Gastrointestinal disorders) | 49 (94)
Oral pain (Gastrointestinal disorders) | 11 (11)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 12 (14)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 38 (60)
Chills (General disorders) | 12 (14)
Edema face (General disorders) | 5 (5)
Edema limbs (General disorders) | 30 (48)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 47 (92)
Fever (General disorders) | 5 (6)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 29 (62)
Injection site reaction (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Neck edema (General disorders) | 3 (4)
Non-cardiac chest pain (General disorders) | 10 (11)
Pain (General disorders) | 15 (17)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (4)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 3 (3)
Immune system disorders - Other, specify (Immune system disorders) | 22 (31)
Appendicitis perforated (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 6 (8)
Enterocolitis infectious (Infections and infestations) | 5 (7)
Infections and infestations - Other, specify (Infections and infestations) | 14 (27)
Lung infection (Infections and infestations) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (5)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 4 (6)
Alanine aminotransferase increased (Investigations) | 44 (78)
Alkaline phosphatase increased (Investigations) | 15 (18)
Aspartate aminotransferase increased (Investigations) | 44 (68)
Blood bilirubin increased (Investigations) | 12 (18)
CPK increased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 5 (5)
Cholesterol high (Investigations) | 4 (4)
Creatinine increased (Investigations) | 12 (18)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Haptoglobin decreased (Investigations) | 1 (1)
INR increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 19 (62)
Lymphocyte count decreased (Investigations) | 52 (104)
Neutrophil count decreased (Investigations) | 51 (100)
Platelet count decreased (Investigations) | 52 (110)
Serum amylase increased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 21 (28)
Weight loss (Investigations) | 14 (17)
White blood cell decreased (Investigations) | 52 (107)
Acidosis (Metabolism and nutrition disorders) | 3 (4)
Alkalosis (Metabolism and nutrition disorders) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 45 (80)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 39 (78)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 10 (11)
Hypernatremia (Metabolism and nutrition disorders) | 7 (7)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 41 (56)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 50 (89)
Hypocalcemia (Metabolism and nutrition disorders) | 36 (58)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 47 (87)
Hypomagnesemia (Metabolism and nutrition disorders) | 48 (73)
Hyponatremia (Metabolism and nutrition disorders) | 47 (79)
Hypophosphatemia (Metabolism and nutrition disorders) | 41 (60)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 19 (86)
Obesity (Metabolism and nutrition disorders) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (35)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (9)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 12 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (34)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7)
Dysgeusia (Nervous system disorders) | 8 (8)
Dysphasia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 40 (65)
Lethargy (Nervous system disorders) | 6 (6)
Memory impairment (Nervous system disorders) | 3 (3)
Movements involuntary (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (8)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (8)
Presyncope (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (2)
Somnolence (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 8 (10)
Agitation (Psychiatric disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 22 (32)
Confusion (Psychiatric disorders) | 12 (14)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 8 (11)
Hallucinations (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 35 (49)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 10 (14)
Psychosis (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 12 (14)
Acute kidney injury (Renal and urinary disorders) | 7 (8)
Hematuria (Renal and urinary disorders) | 10 (11)
Proteinuria (Renal and urinary disorders) | 17 (17)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 14 (17)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 19 (32)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 16 (17)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (13)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (11)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (43)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 34 (42)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 22 (33)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 5 (6)
Hematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 40 (71)
Hypotension (Vascular disorders) | 13 (17)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT01885689/Prot_SAP_000.pdf